CLINICAL TRIAL: NCT04443244
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Phase Ⅱ Optimal Dose-finding Study to Evaluate the Safety and Efficacy of Botulax® in Subjects With Benign Masseteric Hypertrophy
Brief Title: Evaluate the Safety and Efficacy of Botulax® in Subjects With Benign Masseteric Hypertrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HG-BOTBMH-PII-01
Record Dates: First submitted 2020-06-12; First posted 2020-06-23 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Benign Masseteric Hypertrophy
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Botulinum Toxin Type A(Botulax®) 24Units (Experimental): Botulinum Toxin Type A (Botulax®) 24Units total dose administered intramuscularly to the bilateral masseter muscles.
  Interventions: Drug: Botulinum Toxin Type A Injection (Botulax®) 24Units
- Botulinum Toxin Type A(Botulax®) 48Units (Experimental): Botulinum Toxin Type A (Botulax®) 48Units total dose administered intramuscularly to the bilateral masseter muscles.
  Interventions: Drug: Botulinum Toxin Type A Injection (Botulax®) 48Units
- Botulinum Toxin Type A(Botulax®) 72Units (Experimental): Botulinum Toxin Type A (Botulax®) 72Units total dose administered intramuscularly to the bilateral masseter muscles.
  Interventions: Drug: Botulinum Toxin Type A Injection (Botulax®) 72Units
- Botulinum Toxin Type A(Botulax®) 96Units (Experimental): Botulinum Toxin Type A (Botulax®) 96Units total dose administered intramuscularly to the bilateral masseter muscles.
  Interventions: Drug: Botulinum Toxin Type A Injection (Botulax®) 96Units
- Placebo(Normal Saline) (Placebo Comparator): Placebo(Normal saline) administered intramuscularly to the bilateral masseter muscles.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Botulinum Toxin Type A Injection (Botulax®) 24Units — Experimental: Botulax® 24Units
  Other Names: Botulax®
  Arms: Botulinum Toxin Type A(Botulax®) 24Units
Drug: Botulinum Toxin Type A Injection (Botulax®) 48Units — Experimental: Botulax® 48Units
  Other Names: Botulax®
  Arms: Botulinum Toxin Type A(Botulax®) 48Units
Drug: Botulinum Toxin Type A Injection (Botulax®) 72Units — Experimental: Botulax® 72Units
  Other Names: Botulax®
  Arms: Botulinum Toxin Type A(Botulax®) 72Units
Drug: Botulinum Toxin Type A Injection (Botulax®) 96Units — Experimental: Botulax® 96Units
  Other Names: Botulax®
  Arms: Botulinum Toxin Type A(Botulax®) 96Units
Other: Normal Saline — Placebo Comparator: Normal Saline
  Arms: Placebo(Normal Saline)

SUMMARY:
This study is A Randomized, Double-blind, Placebo-controlled, Multi-center Phase II Optimal Dose-finding Study to Evaluate the Safety and Efficacy of Botulax® in Subjects with Benign Masseteric Hypertrophy

DETAILED DESCRIPTION:
A Randomized, Double-blind, Placebo-controlled, Multi-center Phase Ⅱ Optimal Dose-finding Study to Evaluate the Safety and Efficacy of Botulax® in Subjects with Benign Masseteric Hypertrophy

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female adults aged 19 or older.
2. Sighting, facilitation measurement are judged by the investigator to be the ratio of Benign Masseteric Hypertrophy.
3. Subject who understand and willing to perform with the procedures and visiting schedules of clinical trial.
4. Subject who voluntarily agree to participate in this clinical trial.

Exclusion Criteria:

1. Subject who is clinically significant facial asymmetry in visual measurement by the investigator.
2. Fertile women and men who have plans to conceive during pregnancy, breastfeeding and clinical trials or who do not agree to appropriate contraception.
3. Subject who is deemed unable to participate in a clinical trial under the judgement of a Investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Amount of change from baseline in masseter muscle thickness during maximum clenching | Baseline to week 12
  Amount of change from baseline in masseter muscle thickness during maximum clenching by Ultrasonography

SECONDARY OUTCOMES:
Amount of change from baseline in masseter muscle thickness during maximum clenching | Baseline to week 4, 8, 16
  Amount of change from baseline in masseter muscle thickness during maximum clenching by Ultrasonography
Rate of change from baseline in masseter muscle thickness during maximum clenching | Baseline to week 4, 8, 12, 16
  Rate of change from baseline in masseter muscle thickness during maximum clenching by Ultrasonography
Amount of change from baseline in masseter muscle thickness during resting | Baseline to week 4, 8, 12, 16
  Amount of change from baseline in masseter muscle thickness during resting by Ultrasonography
Rate of change from baseline in masseter muscle thickness during resting | Baseline to week 4, 8, 12, 16
  Rate of change from baseline in masseter muscle thickness during resting by Ultrasonography
Amount and rate of change from baseline in lower face volume during maximum clenching | Baseline to week 4, 8, 12, 16
  Amount and rate of change from baseline in lower face volume during maximum clenching by 3D imaging
Overall improvement of Investigator | Baseline to week 4, 8, 12, 16
  Overall improvement of Investigator by assessment scale
Overall satisfaction of subject | Baseline to week 4, 8, 12, 16
  Subject satisfaction assessment using a scale ranging from Extremely dissatisfied to Extremely satisfied by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hugel, Seoul, South Korea